CLINICAL TRIAL: NCT02500693
Title: Circulating Tumor Cells and Early Diagnosis of Lung Cancer in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Circulating Tumor Cells in Lung Cancer Screening
Acronym: AIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-PP-08
Record Dates: First submitted 2015-07-15; First posted 2015-07-16 (Estimated); Last update posted 2024-02-06 (Actual); Status verified 2018-01

CONDITIONS: Lung Neoplasms; Pulmonary Disease, Chronic Obstructive
Keywords: Lung Cancer, Screening, COPD
MeSH Terms: conditions — Lung Neoplasms; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening (Experimental)
  Interventions: Biological: Isolation of circulating tumor cells (CTC) from veinous blood

INTERVENTIONS:
Biological: Isolation of circulating tumor cells (CTC) from veinous blood — Thirty ml of peripheral blood will be collected in buffered EDTA, maintained at 4°C, and processed within 1 hour for filtration. After blood filtration, the membrane will be gently washed with PBS, disassembled from the filtration module, and allowed to air-dry. The determination of CTC number present on filters will be carried out by combining four color immunofluorescent (anti-pancytokeratins/anti-vimentin/DAPI/anti-CD45) staining and cytomorphological examination after Diff-quick and Mayer Hemalun staining in three spots per patient sample. Imaging of immunofluorescent and cytological staining will be performed at x20 magnification using the automated Ariol system. CTCs are identified by relocating images of immunofluorescent and cytological staining.

SUMMARY:
This trial is intended to evaluate the value of circulating tumor cells (CTC), in combination with unenhanced (without injection of contrast media) low dose (to limit the effective radiation dose below 1,5 mSv) chest computed tomography (LDCT) in the screening of Lung cancer (LC).

LDCT screening was shown to reduce LC mortality in smokers and ex-smokers, older than 55 years, with a history of more than 30 pack-years. LDCT however shows a close to 30% rate of false positive that require repeat follow-up and also invasive investigations, but also false negatives with metastatic LC being discovered between screening rounds.

Migration of circulating tumor cells (CTC) is an early event of carcinogenesis and characterizes aggressive cancers. We recently showed that CTC can be detected with the ISET technique in a population at high risk for LC, i.e. COPD patients before LC was detectable on LDCT.

The study will focus on patients at very high risk for lung cancer i.e. smokers and ex-smokers suffering Chronic Obstructive Pulmonary Disease (COPD).

The study will enroll 600 participants who will undergo three rounds of screening at one year intervals, each round combining search for CTC on a blood sample and LDCT. Each participant will be followed for at least one year after the last screening round

ELIGIBILITY:
Inclusion Criteria:

* Age 55 years or more
* 30 or more pack-years of cigarette smoking history
* Former smokers: quit smoking within the previous 15 years
* Signed informed consent form
* Presence of COPD
* Affiliation to the French social security system

Exclusion Criteria:

* Chest CT examination in the 12 months prior to eligibility assessment(1)
* Treatment for, or evidence of, any cancer other than skin basocellular carcinoma in the 5 years prior to eligibility assessment
* Pneumonia or acute respiratory infection treated with antibiotics in the 12 weeks prior to eligibility assessment
* Unexplained weight loss of more than 15 10%pounds in the 12 months prior to eligibility assessment
* Recent hemoptysis
* History of lung volume reduction with coils, glue or valves°
* Metallic implants or devices in the chest or back, such as pacemakers or Harrington fixation rods
* Participation in another cancer screening trial
* Participation in a cancer prevention study, other than a smoking cessation study
* Vulnerable persons: adults under guardianship, adults under trusteeship or persons deprived of their liberty, patients under 18 years old
* Medical and/or psychiatric problems of sufficient severity to limit full compliance with the study or expose patients to undue risk

  1. Many COPD patients will have had a previous chest CT examination. This has become common in medical practice, especially in patients with chronic lung diseases such as COPD patients. Including such patients would introduce huge bias in the study by artificially focusing on rapidly growing cancers. Redoing a CT in a screening intend in a patient who recently underwent this investigation would also unnecessarily enhance irradiation in these patients. It should be note that in the NLST trial "previous chest CT (≤ 18 months)" was a key exclusion criterion [NLST Radiology 2011].

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 683 (Actual)
Dates: Start 2015-10-30 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-13 (Actual)

PRIMARY OUTCOMES:
Rate of detection of circulating tumor cells in patients who will have a LC detected during the study | 3 years

SECONDARY OUTCOMES:
Rate of detection of CTC in the whole study population | once a year for 3 years
Circulating tumor cells | once a year for 3 years
  Predictive value of CTC detection for the diagnosis of LC in patients identified as having a pulmonary nodule.
Time span between detection of CTC and detection of lung cancer with LDCT and vice versa | once a year for 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles-Hugo MARQUETTE, Pr, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (20):
- France (20):
  - CHU d'Amiens, Amiens
  - CHU de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - CHRU de Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - Hôpital Nord, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nancy, Nancy
  - Hôpital Bichat, Paris
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital TENON, Paris
  - CHU de Reims, Reims
  - CHU de Rennes, Rennes
  - CH de Roubaix, Roubaix
  - CHU de Rouen, Rouen
  - CHU de Saint Etienne, Saint-Etienne
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - CHU de Tours, Tours

REFERENCES:
- [Background] Ilie M, Hofman V, Long-Mira E, Selva E, Vignaud JM, Padovani B, Mouroux J, Marquette CH, Hofman P. "Sentinel" circulating tumor cells allow early diagnosis of lung cancer in patients with chronic obstructive pulmonary disease. PLoS One. 2014 Oct 31;9(10):e111597. doi: 10.1371/journal.pone.0111597. eCollection 2014. PMID 25360587
- [Derived] Marquette CH, Boutros J, Benzaquen J, Ferreira M, Pastre J, Pison C, Padovani B, Bettayeb F, Fallet V, Guibert N, Basille D, Ilie M, Hofman V, Hofman P; AIR project Study Group. Circulating tumour cells as a potential biomarker for lung cancer screening: a prospective cohort study. Lancet Respir Med. 2020 Jul;8(7):709-716. doi: 10.1016/S2213-2600(20)30081-3. PMID 32649919
- [Derived] Leroy S, Benzaquen J, Mazzetta A, Marchand-Adam S, Padovani B, Israel-Biet D, Pison C, Chanez P, Cadranel J, Mazieres J, Jounieaux V, Cohen C, Hofman V, Ilie M, Hofman P, Marquette CH; AIR Project Study Group. Circulating tumour cells as a potential screening tool for lung cancer (the AIR study): protocol of a prospective multicentre cohort study in France. BMJ Open. 2017 Dec 26;7(12):e018884. doi: 10.1136/bmjopen-2017-018884. PMID 29282271